CLINICAL TRIAL: NCT01216813
Title: The Rehabilitation Needs of People Who Have Had an Upper Gastrointestinal or a Gynecological Cancer
Brief Title: Study of Physical and Psychosocial Rehabilitation Needs of Patients After Diagnosis and Treatment of Upper Gastrointestinal Cancer or Gynecological Cancer
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000686456; RMNHS-REHABILITATION; EU-21074; RMNHS-CCR3434; MREC-10/H0806/56
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Cervical Cancer; Endometrial Cancer; Esophageal Cancer; Fallopian Tube Cancer; Gastric Cancer; Ovarian Cancer; Sarcoma; Vaginal Cancer; Vulvar Cancer
Keywords: esophageal cancer; gastric cancer; cervical cancer; fallopian tube cancer; ovarian epithelial cancer; ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; endometrial cancer; uterine sarcoma; vaginal cancer; vulvar cancer; adenocarcinoma of the gastroesophageal junction
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Fallopian Tube Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Sarcoma; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Other: informational intervention
Procedure: assessment of therapy complications
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Gathering information from patients who have undergone treatment for upper gastrointestinal cancer or gynecological cancer may help doctors learn more about patients' physical and psychosocial rehabilitation needs and plan the best treatment.

PURPOSE: This clinical trial is studying the physical and psychosocial rehabilitation needs of patients after diagnosis and treatment of upper gastrointestinal cancer or gynecological cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To explore the patients' perspective of their physical and psychosocial rehabilitation needs following the diagnosis and treatment for an upper gastrointestinal or a gynecological cancer.
* To assess patients' experiences of the physical and social impact of cancer in the treatment and post-treatment phase.
* To explore patients' met and un-met needs.
* To explore the patients' opinion of how it might be possible to manage any of the issues that arise.

Secondary

* To generate theories and a hypothesis from the data collected for use in a future interventional study.

OUTLINE: The study consist of a series of focus groups that take place in a private room within the Royal Marsden Hospital in the United Kingdom. Patients attend only one focus group session, which is audio-tape recorded. The focus groups discuss and explore the patient's needs and experiences using a semi-structured interview question schedule over 60-90 minutes. The groups are single-sex groups to allow the patients to express themselves freely with respect to any sensitive topics they may wish to discuss. If individual patient issues arise from the group discussions, the lead researcher may refer the patient to a member of the hospital team, the patient's physician, or for appropriate psychological support.

Data from the focus group dialogue and patients' baseline demographic information are analyzed. The results from this study are used to design an interventional study in the Rehabilitation Department.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of upper gastrointestinal (GI) or gynecological cancer
* Must have completed initial treatment for upper GI or gynecological cancer

  * Received primary treatment within the Royal Marsden NHS Foundation Trust
* Will be on a treatment pathway with radical intent or be post-treatment
* Reported that they have experienced a physical or psychosocial need resulting from the disease or its treatment

PATIENT CHARACTERISTICS:

* Able to attend the specialist center for a focus group session
* Willing and able to articulate their experiences in English
* Not eligible for or receiving palliative or end-of-life care

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Patients' perspective of their physical and psychosocial rehabilitation needs following their diagnosis and treatment
Patients' experiences of the physical and social impact of cancer in the treatment and post-treatment phase
Patients' met and un-met needs
Patients' opinion of how to manage any of the issues that arise

SECONDARY OUTCOMES:
Theories and a hypothesis from data collected for use in a future interventional study

CONTACTS AND LOCATIONS:
Overall Officials: Clare Shaw, Phd, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom